CLINICAL TRIAL: NCT04754932
Title: Implementation of Cognitive Stimulation Therapy Across a Healthcare System to Improve Clinical Outcomes of Individuals Living With Dementing Illnesses
Brief Title: Implementation of Cognitive Stimulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00106751
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Community Site 1 (Experimental): CST Implementation community site
  Interventions: Other: Cognitive Stimulation Therapy
- Community Site 2 (Experimental): CST Implementation community site
  Interventions: Other: Cognitive Stimulation Therapy
- Community Site 3 (Experimental): CST Implementation community site
  Interventions: Other: Cognitive Stimulation Therapy
- Community Site 4 (Experimental): CST Implementation community site
  Interventions: Other: Cognitive Stimulation Therapy
- Community Site 5 (Experimental): CST Implementation community site
  Interventions: Other: Cognitive Stimulation Therapy

INTERVENTIONS:
Other: Cognitive Stimulation Therapy — Group-based therapy for people living with mild to moderate stage dementia, delivered by two trained facilitators.

SUMMARY:
This project aims to examine the feasibility of implementing Cognitive Stimulation Therapy (CST) under real world circumstances in a more heterogenous population, with the ultimate goal of making the treatment broadly accessible. The effects of CST on the behavioral and psychological symptoms of dementia (BPSD) as a non-pharmacologic intervention will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of dementia or meets the criteria for dementia based on a positive screening test with clinical evidence of cognitive impairment affecting one or more ADL
* has a SLUMS score greater than 10.

Exclusion Criteria:

* unable to hold a meaningful conversation,
* unable to hear well enough to participate in a small group discussion
* severe visual impairment that precludes ability to see most pictures
* unable to remain in a group setting for 45 minutes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percent of participants who were eligible for Cognitive Stimulation Therapy but were excluded from participation | 2 years
Change in cognitive status as measured by Saint Louis University Mental Status Examination | Baseline, end-of-protocol (7 weeks), 3-month, 6-month, 12-month
  A validated 30 point office-based cognitive screen
Change in anxiety/depression as measured by Cornell Scale for Depression in Dementia | Baseline, end-of-protocol (7 weeks), 3-month, 6-month, 12-month
  A validated 19 point scale to identify anxiety/depression symptoms in patients with moderate to severe dementia.
Change in quality of life as evaluated by ICEpop CAPability measure for Older people (ICECAP-O) | Baseline, end-of-protocol (7 weeks), 3-month, 6-month, 12-month
  A 5-point scale measuring general well-being/quality of life for older adults
Change in behavioral symptom severity as measured by the Neuropsychiatric Inventory | Baseline, end-of-protocol (7 weeks), 3-month, 6-month, 12-month
  A validated 12-domain questionnaire to assess dementia-related behavioral symptoms
Adoption as measured by the percentage of non-participating centers to the total number approached. | 2 years
Number of CST groups adhering to 18 components of therapy protocol assessed by direct observation using a checklist. | 1 year
Maintenance as measured by percentage of long-term attrition | 2 years
Assess the barriers and facilitators to implementation of CST in community settings | 1 year
  Focus groups will be held to better understand the barriers and facilitators to adoption at both the setting level and individual level. These focus groups will also be used to assess implementation by gathering data on adherence to the prescribed CST protocol and any adaptations made to the CST intervention.
  Implementation fidelity will be assessed by direct observation of the CST groups by members of the research team using a checklist to describe adherence to key components of the protocol. Implementation barriers will be assessed through the use of focus groups and questionnaires. Based on collected data on implementation barriers and process measures, we will develop strategies to improve fidelity of the intervention and to enhance reach.

CONTACTS AND LOCATIONS:
Overall Officials: Milta Little, DO, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Durham Center for Senior Life, Durham, North Carolina
  - Program for All Inclusive Care of the Elderly, Durham, North Carolina
  - The Forest at Duke, Durham, North Carolina
  - Program for All Inclusive Care of the Elderly, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No